CLINICAL TRIAL: NCT06105177
Title: Implementation of Up-front ctDNA Analysis Into Lung Cancer Care and Development of Liquid Biopsy-based Decision Support Models - the Lungmarker² Study
Brief Title: Implementation of Up-front ctDNA Into Lung Cancer Care and Development of Liquid Biopsy-based Decision Support Models - LM² Study
Acronym: LM2
Status: Recruiting | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Eindhoven University of Technology (Other); Roche BV Netherlands (Unknown); Maxima Medical Center (Other); Zuyderland Medisch Centrum (Other); Maastricht University Medical Center (Other); St. Anna Ziekenhuis, Geldrop, Netherlands (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, Volkher Scharnhorst, Prof. Dr. (Clinical Chemist), Catharina Ziekenhuis Eindhoven
Other Study IDs: NL83276.100.22
Record Dates: First submitted 2023-10-17; First posted 2023-10-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
Keywords: lungmarker2 study; lung cancer; liquid biopsy; ctDNA; CTCs; tumormarkers
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — * Whole blood drawn into serum tubes for the measurement of tumormarkers (CA125, CA15.3, CEA, CYFRA 21.1, HE-4, NSE, proGRP, SCCA)
  * Whole blood drawn into cell preservation tubes for ctDNA analysis and isolation of circulating tumor cells (CTCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite scientific evidence, use of liquid biopsy (LB) in diagnosis and monitoring of lung cancer (LC) is limited since it requires major changes in diagnostic and care pathways. Analyzing tumor markers (TMs), circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA) in blood (LB) can inform about the nature of the tumor, the most appropriate therapy, therapy response and resistance.

Lungmarker2 is a multicenter, prospective, implementation and diagnostic cohort study. This study aims to implement up-front ctDNA analysis ('plasma first approach') into routine diagnostic work-up of all advanced stage LC patients in the Southeast of the Netherlands (the participating hospitals in the OncoZON region). Thereby, additional information about the molecular make-up of the tumor becomes available, the number of tissue Next-Generation Sequencing (NGS) analyses will decrease and time to therapeutic decision making is shortened. Next, using ctDNA, TM and other information, multi-parametric decision support models are built and validated that may support diagnosis, predict the outcome of the next imaging procedure and progression-free survival during follow-up. The final goal is to develop a super-resolution microscopy test that can detect PD-L1 expression on CTCs.

DETAILED DESCRIPTION:
RATIONALE: Despite scientific evidence, use of liquid biopsy (LB) in diagnosis and monitoring of lung cancer (LC) is limited since it requires major changes in diagnostic and care pathways. Analyzing tumor markers (TMs), circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA) in blood (LB) can inform about the nature of the tumor, the most appropriate therapy, therapy response and resistance.

OBJECTIVE: To implement up-front ctDNA analysis ('plasma first approach') into routine diagnostic work-up of all advanced stage LC patients in the Southeast of the Netherlands (the participating hospitals in the OncoZON region) and to thereby validate that significantly more information about the molecular make-up of the tumor becomes available by introduction of up-front ctDNA. To establish that the number of tissue NGS analyses decreases and time to therapeutic decision making is shortened. To build and to validate, using ctDNA, TM and other information, multiparametric decision support models that may support diagnosis, predict the outcome of the next imaging procedure and survival during follow up. The final goal is to develop a super-resolution microscopy test that can detect PD-L1 expression on CTCs.

STUDY DESIGN: Multicenter, prospective, implementation and diagnostic cohort study.

STUDY POPULATION: 800 patients suspected of having lung cancer.

MAIN STUDY PARAMETERS/ENDPOINTS: ctDNA analysis, as additional source of genetic information, has been integrated into the diagnostic workup of LC patients and the medical benefits thereof are quantified, e.g. a significant higher percentage of patients with a driver mutation is identified by introduction of the plasma first approach. Multiparametric decision support algorithms based on imaging, TM and ctDNA analyses that identify small-cell LC (SCLC) and non-small-cell LC (NSCLC) have been developed and validated. Multiparametric decision support models have been developed that enable patient-specific timing of imaging procedures and predict survival during follow-up of LC patients. A super-resolution microscopy test for PD-L1 is developed and correlation with tumor tissue PD-L1 expression has been established.

NATURE AND EXTENT OF THE BURDEN AND RISKS ASSOCIATED WITH PARTICIPATION, BENEFIT AND GROUP RELATEDNESS: At diagnosis, an extra 10 mL of blood are drawn during a routine venipuncture. Patients with advanced stage LC (stage IIIb/c or IV) undergo an extra venipuncture (40 mL).The longest follow up period for a patient is 36 months with a maximum of 20 blood draws. The volume per draw ranges from 10-40 mL. The risks of a venipuncture are negligible and the burden minimal. Those patients for whom a targetable mutation is found by ctDNA analysis benefit from the advantages of targeted therapy, i.e. better survival and less side effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above and suspected of having lung cancer

Exclusion Criteria:

* Presence of another malignant tumor, i.e. diagnosed with a tumor in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 800 individuals, >18 years of age, suspected of lung cancer and referred to a lung physician in one of the participating centers are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Up-front ctDNA analysis is implemented into routine clinical care in the participating OncoZoN hospitals | Up to 3 years
  After the Lungmarker2 study has proven up-front ctDNA analysis to be feasible and successful for diagnosis and monitoring of lung cancer, hospitals participating in this project will adopt this as routine practice. Up-front ctDNA analysis will be adopted by the other OncoZON hospitals outside the consortium through transfer of the clinical practice during the regular tumor board meetings where shared care decisions are made for individual patients.
Evaluate the number of driver mutations detected by up-front ctDNA analysis compared to tumor NGS analysis | Up to 3 years
  Determine and compare the number of driver mutations detected by up-front ctDNA analysis with the number of driver mutations detected by tumor NGS analysis.
Develop decision support algorithms for the diagnosis and monitoring of lung cancer patients | Up to 3 years
  Develop decision support algorithms using information from CT scans, measured tumor markers (CA125, CA15.3, CEA, CYFRA 21.1, HE-4, NSE, proGRP, SCCA) and ctDNA analysis to identify small-cell lung cancer and non-small-cell lung cancer patients (classification, diagnosis).
  Develop decision support algorithms to predict therapy response, expressed as a threshold for durable clinical benefit: the progression free survival (PFS) at 6 months (as probability %), in lung cancer patients (monitoring).
  Different metrics regarding model performances will be reported: area under the receiver operating characteristic curve (AUC), area under the precision- recall curve (AUC-PR), sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV).

SECONDARY OUTCOMES:
Develop an analytical protocol for the analysis of PD-L1 expression on circulating tumor cells (CTCs) by super-resolution microscopy | Up to 3 years
  Develop an analytical protocol for the isolation of CTCs from whole blood samples (measured as the number of cells per mL) and to quantify PD-L1 expression (reported as a percentage on a scale of 0% to 100%) on the isolated CTCs using super-resolution microscopy.
Evaluate the number of tumor NGS analyses and time to diagnosis when up-front ctDNA analysis is introduced | Up to 3 years
  Determine the time to diagnosis (in days) of lung cancer (e.g., time between first visit at lung physician and the diagnosis) when using up-front ctDNA analysis compared to tumor NGS analysis, and determine the number of tumor NGS analyses that can be replaced by up-front ctDNA analysis.

OTHER OUTCOMES:
A study database is filled with all relevant clinical and diagnostic information | Up to 3 years
  For the Lungmarker2 study, all information will be entered into the study database (Research manager) by personnel of the participating hospitals (research nurse, physician or lung oncology nurse) using a digital CRF. Research manager offers eCRF possibilities and enables safe and anonymous data collection, storage and management. The data collected include patient data, detailed results of diagnostic procedures and tests including imaging procedures, treatment regime and response evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Volkher Scharnhorst, Prof.Dr., Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (5):
- Netherlands (5):
  - Zuyderland Medical Center, Heerlen, Limburg
  - Maastricht University Medical Center, Maastricht, Limburg
  - Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant
  - St. Anna Ziekenhuis, Geldrop, North Brabant
  - Máxima Medisch Centrum, Veldhoven, North Brabant

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ignatiadis M, Sledge GW, Jeffrey SS. Liquid biopsy enters the clinic - implementation issues and future challenges. Nat Rev Clin Oncol. 2021 May;18(5):297-312. doi: 10.1038/s41571-020-00457-x. Epub 2021 Jan 20. PMID 33473219
- [Background] IJzerman MJ, de Boer J, Azad A, Degeling K, Geoghegan J, Hewitt C, Hollande F, Lee B, To YH, Tothill RW, Wright G, Tie J, Dawson SJ. Towards Routine Implementation of Liquid Biopsies in Cancer Management: It Is Always Too Early, until Suddenly It Is Too Late. Diagnostics (Basel). 2021 Jan 11;11(1):103. doi: 10.3390/diagnostics11010103. PMID 33440749
- [Background] Rolfo C, Mack P, Scagliotti GV, Aggarwal C, Arcila ME, Barlesi F, Bivona T, Diehn M, Dive C, Dziadziuszko R, Leighl N, Malapelle U, Mok T, Peled N, Raez LE, Sequist L, Sholl L, Swanton C, Abbosh C, Tan D, Wakelee H, Wistuba I, Bunn R, Freeman-Daily J, Wynes M, Belani C, Mitsudomi T, Gandara D. Liquid Biopsy for Advanced NSCLC: A Consensus Statement From the International Association for the Study of Lung Cancer. J Thorac Oncol. 2021 Oct;16(10):1647-1662. doi: 10.1016/j.jtho.2021.06.017. Epub 2021 Jul 8. PMID 34246791
- [Background] de Kock R, Deiman B, Kraaijvanger R, Scharnhorst V. Optimized (Pre) Analytical Conditions and Workflow for Droplet Digital PCR Analysis of Cell-Free DNA from Patients with Suspected Lung Carcinoma. J Mol Diagn. 2019 Sep;21(5):895-902. doi: 10.1016/j.jmoldx.2019.05.003. Epub 2019 Jun 21. PMID 31229652
- [Background] Genet SAAM, Visser E, van den Borne BEEM, Soud MY, Belderbos HNA, Stege G, de Saegher MEA, Eduati F, Broeren MAC, van Dongen J, Brunsveld L, van de Kerkhof D, Scharnhorst V. Correction of the NSE concentration in hemolyzed serum samples improves its diagnostic accuracy in small-cell lung cancer. Oncotarget. 2020 Jul 7;11(27):2660-2668. doi: 10.18632/oncotarget.27664. eCollection 2020 Jul 7. PMID 32676167
- [Background] de Kock R, van den Borne B, Youssef-El Soud M, Belderbos H, Brunsveld L, Scharnhorst V, Deiman B. Therapy Monitoring of EGFR-Positive Non-Small-Cell Lung Cancer Patients Using ddPCR Multiplex Assays. J Mol Diagn. 2021 Apr;23(4):495-505. doi: 10.1016/j.jmoldx.2021.01.003. Epub 2021 Jan 22. PMID 33486072
- [Background] de Kock R, Knoops C, Baselmans M, Borne BVD, Brunsveld L, Scharnhorst V, Deiman B. Sensitive cell-free tumor DNA analysis in supernatant pleural effusions supports therapy selection and disease monitoring of lung cancer patients. Cancer Treat Res Commun. 2021;29:100449. doi: 10.1016/j.ctarc.2021.100449. Epub 2021 Aug 25. PMID 34481168
- [Background] de Kock R, Borne BVD, Soud MY, Belderbos H, Stege G, de Saegher M, van Dongen-Schrover C, Genet S, Brunsveld L, Scharnhorst V, Deiman B. Circulating biomarkers for monitoring therapy response and detection of disease progression in lung cancer patients. Cancer Treat Res Commun. 2021;28:100410. doi: 10.1016/j.ctarc.2021.100410. Epub 2021 Jun 1. PMID 34107412
- [Background] Visser E, de Kock R, Genet S, Borne BVD, Soud MY, Belderbos H, Stege G, de Saegher M, 't Westeinde SV, Broeren M, Eduati F, Deiman B, Scharnhorst V. Up-front mutation detection in circulating tumor DNA by droplet digital PCR has added diagnostic value in lung cancer. Transl Oncol. 2023 Jan;27:101589. doi: 10.1016/j.tranon.2022.101589. Epub 2022 Nov 19. PMID 36413862
- [Background] Visser E, Genet SAAM, de Kock RPPA, van den Borne BEEM, Youssef-El Soud M, Belderbos HNA, Stege G, de Saegher MEA, van 't Westeinde SC, Brunsveld L, Broeren MAC, van de Kerkhof D, Deiman BALM, Eduati F, Scharnhorst V. Liquid biopsy-based decision support algorithms for diagnosis and subtyping of lung cancer. Lung Cancer. 2023 Apr;178:28-36. doi: 10.1016/j.lungcan.2023.01.014. Epub 2023 Feb 1. PMID 36773458
- [Background] Hendriks LE, Kerr KM, Menis J, Mok TS, Nestle U, Passaro A, Peters S, Planchard D, Smit EF, Solomon BJ, Veronesi G, Reck M; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Oncogene-addicted metastatic non-small-cell lung cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2023 Apr;34(4):339-357. doi: 10.1016/j.annonc.2022.12.009. Epub 2023 Jan 23. No abstract available. PMID 36872130
- [Background] Hendriks LE, Kerr KM, Menis J, Mok TS, Nestle U, Passaro A, Peters S, Planchard D, Smit EF, Solomon BJ, Veronesi G, Reck M; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Non-oncogene-addicted metastatic non-small-cell lung cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2023 Apr;34(4):358-376. doi: 10.1016/j.annonc.2022.12.013. Epub 2023 Jan 17. No abstract available. PMID 36669645
- [Background] Finall A, Davies G, Jones T, Emlyn G, Huey P, Mullard A. Integration of rapid PCR testing as an adjunct to NGS in diagnostic pathology services within the UK: evidence from a case series of non-squamous, non-small cell lung cancer (NSCLC) patients with follow-up. J Clin Pathol. 2023 Jun;76(6):391-399. doi: 10.1136/jclinpath-2021-207987. Epub 2022 Jan 18. PMID 35042754
- [Background] Thompson JC, Aggarwal C, Wong J, Nimgaonkar V, Hwang WT, Andronov M, Dibardino DM, Hutchinson CT, Ma KC, Lanfranco A, Moon E, Haas AR, Singh AP, Ciunci CA, Marmarelis M, D'Avella C, Cohen JV, Bauml JM, Cohen RB, Langer CJ, Vachani A, Carpenter EL. Plasma Genotyping at the Time of Diagnostic Tissue Biopsy Decreases Time-to-Treatment in Patients With Advanced NSCLC-Results From a Prospective Pilot Study. JTO Clin Res Rep. 2022 Mar 8;3(4):100301. doi: 10.1016/j.jtocrr.2022.100301. eCollection 2022 Apr. PMID 35392653
- [Background] Hendriks LEL, Dingemans AC, De Ruysscher DKM, Aarts MJ, Barberio L, Cornelissen R, Hartemink KJ, van den Heuvel M, Schuuring E, Smit HJM, van der Wekken AJ, Smit EF. Lung Cancer in the Netherlands. J Thorac Oncol. 2021 Mar;16(3):355-365. doi: 10.1016/j.jtho.2020.10.012. No abstract available. PMID 33641718
- [Background] Imamura F, Uchida J, Kukita Y, Kumagai T, Nishino K, Inoue T, Kimura M, Kato K. Early responses of EGFR circulating tumor DNA to EGFR tyrosine kinase inhibitors in lung cancer treatment. Oncotarget. 2016 Nov 1;7(44):71782-71789. doi: 10.18632/oncotarget.12373. PMID 27708242
- [Background] Goldberg SB, Narayan A, Kole AJ, Decker RH, Teysir J, Carriero NJ, Lee A, Nemati R, Nath SK, Mane SM, Deng Y, Sukumar N, Zelterman D, Boffa DJ, Politi K, Gettinger SN, Wilson LD, Herbst RS, Patel AA. Early Assessment of Lung Cancer Immunotherapy Response via Circulating Tumor DNA. Clin Cancer Res. 2018 Apr 15;24(8):1872-1880. doi: 10.1158/1078-0432.CCR-17-1341. Epub 2018 Jan 12. PMID 29330207
- [Background] Di Capua D, Bracken-Clarke D, Ronan K, Baird AM, Finn S. The Liquid Biopsy for Lung Cancer: State of the Art, Limitations and Future Developments. Cancers (Basel). 2021 Aug 4;13(16):3923. doi: 10.3390/cancers13163923. PMID 34439082
- [Background] Honrubia-Peris B, Garde-Noguera J, Garcia-Sanchez J, Piera-Molons N, Llombart-Cussac A, Fernandez-Murga ML. Soluble Biomarkers with Prognostic and Predictive Value in Advanced Non-Small Cell Lung Cancer Treated with Immunotherapy. Cancers (Basel). 2021 Aug 25;13(17):4280. doi: 10.3390/cancers13174280. PMID 34503087
- [Background] Molina R, Marrades RM, Auge JM, Escudero JM, Vinolas N, Reguart N, Ramirez J, Filella X, Molins L, Agusti A. Assessment of a Combined Panel of Six Serum Tumor Markers for Lung Cancer. Am J Respir Crit Care Med. 2016 Feb 15;193(4):427-37. doi: 10.1164/rccm.201404-0603OC. PMID 26465739
- [Background] Olmedillas-Lopez S, Garcia-Arranz M, Garcia-Olmo D. Current and Emerging Applications of Droplet Digital PCR in Oncology. Mol Diagn Ther. 2017 Oct;21(5):493-510. doi: 10.1007/s40291-017-0278-8. PMID 28477149
- [Background] Schouten RD, Vessies DCL, Bosch LJW, Barlo NP, van Lindert ASR, Cillessen SAGM, van den Broek D, van den Heuvel MM, Monkhorst K. Clinical Utility of Plasma-Based Comprehensive Molecular Profiling in Advanced Non-Small-Cell Lung Cancer. JCO Precis Oncol. 2021 Jul 9;5:PO.20.00450. doi: 10.1200/PO.20.00450. eCollection 2021 Jul. PMID 34632253
- [Background] van den Broek D, Hiltermann TJN, Biesma B, Dinjens WNM, 't Hart NA, Hinrichs JWJ, Leers MPG, Monkhorst K, van Oosterhout M, Scharnhorst V, Schuuring E, Speel EM, van den Heuvel MM, van Schaik RHN, von der Thusen J, Willems SM, de Visser L, Ligtenberg MJL. Implementation of Novel Molecular Biomarkers for Non-small Cell Lung Cancer in the Netherlands: How to Deal With Increasing Complexity. Front Oncol. 2020 Jan 22;9:1521. doi: 10.3389/fonc.2019.01521. eCollection 2019. PMID 32039011
- [Background] Moritz R, Muller M, Korse CM, van den Broek D, Baas P, van den Noort V, Ten Hoeve JJ, van den Heuvel MM, van Rossum HH. Diagnostic validation and interpretation of longitudinal circulating biomarkers using a biomarker response characteristic plot. Clin Chim Acta. 2018 Dec;487:6-14. doi: 10.1016/j.cca.2018.09.015. Epub 2018 Sep 8. PMID 30201371
- [Background] Verheijen RB, van Duijl TT, van den Heuvel MM, Vessies D, Muller M, Beijnen JH, Janssen JM, Schellens JHM, Steeghs N, van den Broek D, Huitema ADR. Monitoring of EGFR mutations in circulating tumor DNA of non-small cell lung cancer patients treated with EGFR inhibitors. Cancer Chemother Pharmacol. 2021 Feb;87(2):269-276. doi: 10.1007/s00280-021-04230-4. Epub 2021 Jan 23. PMID 33484280
- [Background] Cisneros-Villanueva M, Hidalgo-Perez L, Rios-Romero M, Cedro-Tanda A, Ruiz-Villavicencio CA, Page K, Hastings R, Fernandez-Garcia D, Allsopp R, Fonseca-Montano MA, Jimenez-Morales S, Padilla-Palma V, Shaw JA, Hidalgo-Miranda A. Cell-free DNA analysis in current cancer clinical trials: a review. Br J Cancer. 2022 Feb;126(3):391-400. doi: 10.1038/s41416-021-01696-0. Epub 2022 Jan 13. PMID 35027672
- [Background] Nabet BY, Esfahani MS, Moding EJ, Hamilton EG, Chabon JJ, Rizvi H, Steen CB, Chaudhuri AA, Liu CL, Hui AB, Almanza D, Stehr H, Gojenola L, Bonilla RF, Jin MC, Jeon YJ, Tseng D, Liu C, Merghoub T, Neal JW, Wakelee HA, Padda SK, Ramchandran KJ, Das M, Plodkowski AJ, Yoo C, Chen EL, Ko RB, Newman AM, Hellmann MD, Alizadeh AA, Diehn M. Noninvasive Early Identification of Therapeutic Benefit from Immune Checkpoint Inhibition. Cell. 2020 Oct 15;183(2):363-376.e13. doi: 10.1016/j.cell.2020.09.001. Epub 2020 Oct 1. PMID 33007267
- [Background] Julie Horrocks. Marianne J. van Den Heuvel.
- [Background] Ibrahim JG, Chu H, Chen LM. Basic concepts and methods for joint models of longitudinal and survival data. J Clin Oncol. 2010 Jun 1;28(16):2796-801. doi: 10.1200/JCO.2009.25.0654. Epub 2010 May 3. PMID 20439643
- [Background] Schermelleh L, Ferrand A, Huser T, Eggeling C, Sauer M, Biehlmaier O, Drummen GPC. Super-resolution microscopy demystified. Nat Cell Biol. 2019 Jan;21(1):72-84. doi: 10.1038/s41556-018-0251-8. Epub 2019 Jan 2. PMID 30602772
- [Background] Winckler P, Lartigue L, Giannone G, De Giorgi F, Ichas F, Sibarita JB, Lounis B, Cognet L. Identification and super-resolution imaging of ligand-activated receptor dimers in live cells. Sci Rep. 2013;3:2387. doi: 10.1038/srep02387. PMID 23925048
- [Background] Riera R, Hogervorst TP, Doelman W, Ni Y, Pujals S, Bolli E, Codee JDC, van Kasteren SI, Albertazzi L. Single-molecule imaging of glycan-lectin interactions on cells with Glyco-PAINT. Nat Chem Biol. 2021 Dec;17(12):1281-1288. doi: 10.1038/s41589-021-00896-2. Epub 2021 Nov 11. PMID 34764473
- [Background] Delcanale P, Porciani D, Pujals S, Jurkevich A, Chetrusca A, Tawiah KD, Burke DH, Albertazzi L. Aptamers with Tunable Affinity Enable Single-Molecule Tracking and Localization of Membrane Receptors on Living Cancer Cells. Angew Chem Int Ed Engl. 2020 Oct 12;59(42):18546-18555. doi: 10.1002/anie.202004764. Epub 2020 Aug 28. PMID 32627326
- [Background] Schnitzbauer J, Strauss MT, Schlichthaerle T, Schueder F, Jungmann R. Super-resolution microscopy with DNA-PAINT. Nat Protoc. 2017 Jun;12(6):1198-1228. doi: 10.1038/nprot.2017.024. Epub 2017 May 18. PMID 28518172
- [Background] Shen H, Tauzin LJ, Baiyasi R, Wang W, Moringo N, Shuang B, Landes CF. Single Particle Tracking: From Theory to Biophysical Applications. Chem Rev. 2017 Jun 14;117(11):7331-7376. doi: 10.1021/acs.chemrev.6b00815. Epub 2017 May 18. PMID 28520419
- See also: de Kock RPPAW. Tumor markers in diagnosis and therapy monitoring of lung cancer. Technische Universiteit Eindhoven; 2021. — https://pure.tue.nl/ws/portalfiles/portal/190681670/20211214_Kock.pdf